CLINICAL TRIAL: NCT02184949
Title: Percutaneous Coronary Interventions in the UK: The Relationship Between Procedural Volumes and Patient Outcomes in a Changing Context (A NICOR Study)
Brief Title: Exploring the Volume-Outcome Relationship for PCI Procedures Undertaken in a UK Context: A NICOR Study
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: National Institute for Cardiovascular Outcomes Research (Other); British Cardiovascular Society (Unknown); British Cardiovascular Intervention Society (Other)
Responsible Party: Principal Investigator, Dara O'Neill, Information Analyst, University College, London
Other Study IDs: NICOR-PCI-VolOut
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Percutaneous Coronary Intervention
Keywords: PCI; Coronary angioplasty; Percutaneous transluminal coronary angioplasty; PTCA
MeSH Terms: interventions — Percutaneous Coronary Intervention; Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Sample: All percutaneous coronary intervention patients who meet the primary eligibility criteria for this study.
  Interventions: Procedure: Percutaneous Coronary Intervention
- Subsample: Patients drawn from the main sample who specifically underwent a primary percutaneous coronary intervention procedure.
  Interventions: Procedure: Primary Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention
  Other Names: PCI; Coronary angioplasty
  Groups: Primary Sample
Procedure: Primary Percutaneous Coronary Intervention
  Other Names: pPCI; Primary angioplasty
  Groups: Subsample

SUMMARY:
The relationship between annual procedural volume and patient outcome remains a debated issue in the field of interventional medicine. An under-explored issue in a UK context is whether or not such a relationship exists for percutaneous coronary interventions (PCI). In recent years, this procedure has replaced thrombolysis as the standard intervention method used in UK hospitals for widening patients' obstructed coronary arteries. However, the actual number of such procedures currently undertaken annually remains variable across hospitals where these interventions are performed. The UK's National Institute for Health and Care Excellence has consequently called for research into whether such differences in volume play any role in patient outcome for this particular procedure. The current study is intended to address that research need, and will do so by looking at whether the annual number of PCI procedures undertaken by individual hospitals is predictive of patient mortality post-procedure.

DETAILED DESCRIPTION:
Using data collected as part of a UK national audit of percutaneous coronary interventions, this study will:

* Establish whether annual hospital volume is a clinically important novel risk factor for 30-day mortality post-PCI when examined relative to a newly developed risk model intended for use in clinical practice.
* Establish whether the nature of this volume-outcome relationship is best fit as a linear or non-linear model.
* Establish whether annual hospital volume is a clinically important novel risk factor for 30-day mortality post-primary PCI when examined relative to a newly developed risk model intended for use in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* are aged between 18 and 100 (inclusive) on the date of their procedure;
* do not have pre-operative ventilation;
* undergo a PCI procedure in a UK hospital that contributes data to the National Audit of Percutaneous Coronary Intervention; and
* have a tracked mortality status at 30 days' post-procedure.

To account for potential dependencies in the data, patients' non-index (i.e. follow-up) PCI procedures occurring during the data collection period will be excluded from the study sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Percutaneous coronary interventions undertaken in UK hospitals are recorded in the UK National Audit of Percutaneous Coronary Intervention. Patients who contribute data to this audit will be eligible for inclusion in this study. Additional inclusion criteria, as described below, will be applied to ensure that data are appropriate for the intended analysis.
Sampling Method: Non-Probability Sample
Enrollment: 427467 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: D O'Neill, PhD, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

REFERENCES:
- [Derived] O'Neill D, Nicholas O, Gale CP, Ludman P, de Belder MA, Timmis A, Fox KA, Simpson IA, Redwood S, Ray SG. Total Center Percutaneous Coronary Intervention Volume and 30-Day Mortality: A Contemporary National Cohort Study of 427 467 Elective, Urgent, and Emergency Cases. Circ Cardiovasc Qual Outcomes. 2017 Mar;10(3):e003186. doi: 10.1161/CIRCOUTCOMES.116.003186. PMID 28320707